CLINICAL TRIAL: NCT01576133
Title: Reducing Disability Via a Bundled Bio-Behavioral-Environmental Approach
Acronym: CAPABLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NA_00031539; R01AG040100 (NIH)
Record Dates: First submitted 2012-04-04; First posted 2012-04-12 (Estimated); Last update posted 2018-07-02 (Actual); Status verified 2018-06

CONDITIONS: Quality of Life
Keywords: Quality of Life
MeSH Terms: interventions — CAPABLE protocol

STUDY DESIGN:
Intervention Model Description: Time limited home based intervention of a Nurse, Occupational Therapist, and a "handyman" to work with low income older adults to assess, prioritize and meet their functional goals.
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor did not know which study group the person they visited was in and told participant not to reveal it.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CAPABLE (Experimental): Experimental group participants received up to 10 sessions; up to 6 with an OT, and up to 4 sessions with an RN, and ≤ $1200 of safety and functional modifications from a licensed handyman. These sessions happened in coordinated fashion over the course of 4 months.
  Interventions: Behavioral: CAPABLE
- Attention visits (Active Comparator): Participants in the attention visit arm received 10 visits of one hour length spaced across 16 weeks. These visits included sedentary activities of their choice based on their goals and interests.
  Interventions: Behavioral: Attention visits

INTERVENTIONS:
Behavioral: CAPABLE — Occupational therapy visits plus nursing visits plus handyman repair
  Arms: CAPABLE
Behavioral: Attention visits — Participants in the attention control arm will receive 10 one hour visits over the course of 16 weeks. These visits will consist of sedentary activities
  Arms: Attention visits

SUMMARY:
The purpose of the study is to determine whether a combination of occupational therapy visits, nursing visits, and handyman repair are effective in helping low income older adults avoid costly health care services

DETAILED DESCRIPTION:
We will recruit low-income age 65 or older

-principally African-American, adults from the Baltimore Department of Housing Energy Assistance Program.

-We will interview them at home and randomize participants to either the treatment (CAPABLE intervention) or control (attention-control) group. Participants in the treatment group will receive up to 10 in-home sessions -- 6 visits with an occupational therapist and 4 visits from a nurse - and $1200 in safety and modification services from a licensed handyman. Each treatment participant will receive each intervention component but interventionists will systematically tailor content to the participants' risk profile and goals based on protocols.

ELIGIBILITY:
Inclusion Criteria:

* at least 65 years old
* cognitively intact
* difficulty with at least one activity of daily living or two instrumental activities of daily living
* less than 175% of the Federal Poverty level
* be able to stand with or without assistance
* agree to study participation

Exclusion Criteria:

* hospitalized more than three times in the last year
* receiving in home rehabilitation
* have a terminal diagnosis with less than one year life expectancy
* plan to move in less than one year

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 300 (Actual)
Dates: Start 2012-04; Primary Completion 2017-04 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Activities of Daily Living (ADLs) | 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Szanton, PhD, ANP, Principal Investigator — Johns Hopkins University School of Nursing
Locations (1):
- Johns Hopkins University School of Nursing, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Szanton SL, Xue QL, Leff B, Guralnik J, Wolff JL, Tanner EK, Boyd C, Thorpe RJ Jr, Bishai D, Gitlin LN. Effect of a Biobehavioral Environmental Approach on Disability Among Low-Income Older Adults: A Randomized Clinical Trial. JAMA Intern Med. 2019 Feb 1;179(2):204-211. doi: 10.1001/jamainternmed.2018.6026. PMID 30615024
- [Derived] Waldersen BW, Wolff JL, Roberts L, Bridges AE, Gitlin LN, Szanton SL. Functional Goals and Predictors of Their Attainment in Low-Income Community-Dwelling Older Adults. Arch Phys Med Rehabil. 2017 May;98(5):896-903. doi: 10.1016/j.apmr.2016.11.017. Epub 2016 Dec 19. PMID 28007445